CLINICAL TRIAL: NCT05954702
Title: Supercharged TRAM Evaluation in Cervical Esophagogastroplasty After Esophagectomy
Acronym: Supercharged
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NP 1683
Record Dates: First submitted 2023-06-30; First posted 2023-07-20 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-06

CONDITIONS: Esophagus Cancer; Carcinoma Esophagus
Keywords: Esophagectomy; Esophagogastroplasty; Supercharged
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Esophagectomy group (Active Comparator): Patients with malignant esophagus neoplasms randomized to Conventional Esophagectomy will undergo to an esophagectomy, immediately followed by an esophagus reconstruction trough esophagogastroplasty.
  Interventions: Procedure: Conventional Esophagectomy
- Supercharged TRAM esophagectomy group (Experimental): Patients with malignant esophagus neoplasms randomized to Supercharged TRAM esophagectomy will undergo to esophagectomy, immediately followed by supercharged esophagogastroplasty.
  Interventions: Procedure: Supercharged TRAM esophagectomy

INTERVENTIONS:
Procedure: Supercharged TRAM esophagectomy — Esophagectomy, immediately followed by supercharged esophagogastroplasty. Use the transverse rectus abdominis myocutaneous (TRAM) flap transfers to surgically create a new anastomosis in the left gastroepiploic vessels.
  Arms: Supercharged TRAM esophagectomy group
Procedure: Conventional Esophagectomy — Esophagectomy, immediately followed by an esophagus reconstruction trough esophagogastroplasty.
  Arms: Conventional Esophagectomy group

SUMMARY:
Esophagectomy has high rates of morbidity and mortality, in many cases due to esophagus reconstruction. Anastomotic leakage and fistula are the main esophagectomy complications. Many studies underwent to investigate the cause for anastomotic leakage after esophagectomy, however none of them conclude it is related to surgery or suture technique. However, it seems to be triggered by the ischemia caused after stomach mobilization to esophagus reconstruction, or even tension in the anastomosis.

Considering the post esophagectomy with gastroplasty high morbidity and mortality rates, strategies to create a new vascularization source and decrease anastomotic leakage rates is important. In this study researchers will evaluate whether a TRAM flap transfer supercharged is effective on decrease morbidity related to anastomosis ischemia in patients undergoing esophagectomy.

DETAILED DESCRIPTION:
The transfer of muscle parts is one of the main reconstruction techniques used in plastic surgery. Transverse rectus abdominis myocutaneous (TRAM) flap transfers are very considered due to high quality results, wide application in many cases, and small number of reviews in long term.

Beegle, in 1991 published a new technique of using TRAM supercharged in which microsurgical anastomosis are used between TRAM's unipedicled gastroepiploic deep artery and veins and thoracic branches and vessels, such as axillary and thoracodorsal vessels.

Looking for recover tissue blood perfusion and decrease morbidity rates associated with anastomosis ischemia, some studies showed large intestine or jejunum interposition plus an additional blood supply through venous and arterial anastomosis - colon or jejunum supercharged is effective. The isoperistaltic supercharged colon interposition was a good option to rebuild big esophagus parts in which stomach was not available.

Considering the post esophagectomy with gastroplasty high morbidity and mortality rates, strategies to create a new vascularization source and decrease anastomotic leakage rates is important. This is a single-institution, randomized clinical trial with participants recruited in the digestive system surgery clinic, at the Instituto do Câncer do Estado de São Paulo (ICESP). Patients will be randomized to conventional esophagectomy or TRAM supercharged esophagectomy, and researchers will evaluate post-operatory complications in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of esophageal malignancy cancer;
* Ability to understand and collaborate during treatment;

Exclusion Criteria:

* Previous gastrectomy;
* Previous abdominal surgery with risk of altering stomach vascularization;
* Previous head and neck surgery with risk of alteration of cervical vessels.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-21 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Presence and number of post-operatory complications | Until 1 year after Surgery
  surgical wound infection, hematoma, anastomotic leakage, stenosis, chylothorax and clinical complications due to hospitalization
Mortality | Until 1 year after surgery after surgery
  Patients who and when died

SECONDARY OUTCOMES:
Days in intensive care unit | From the surgery day until the date patient leave intensive care unit
  Number of days patient will stay at intensive care unit
Hospitalization period | From the surgery day until the date patient leave hospital
  Number of days patient will stay in hospital after surgery
Need of vasoactive drugs | From the surgery day until the date patient leave hospital
  If patient use vasoactive drugs drugs hospitalization
Blood transfusion need | From the surgery day until the date patient leave hospital
  If patients need blood transfusion during hospitalization
Drain use time | From the surgery day until the date patient took off drain
  How long patient use drain

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Takeda, PhD, MD, Principal Investigator — Instituto do Cancer do Estado de São Paulo
Locations (1):
- Instituto do Cancer do Estado de São Paulo (ICESP), São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akiyama H. Surgery for carcinoma of the esophagus. Curr Probl Surg. 1980 Feb;17(2):53-120. doi: 10.1016/s0011-3840(80)80025-6. No abstract available. PMID 6987040
- [Background] Akiyama H, Miyazono H, Tsurumaru M, Hashimoto C, Kawamura T. Use of the stomach as an esophageal substitute. Ann Surg. 1978 Nov;188(5):606-10. doi: 10.1097/00000658-197811000-00004. PMID 718285
- [Background] Barzin A, Norton JA, Whyte R, Lee GK. Supercharged jejunum flap for total esophageal reconstruction: single-surgeon 3-year experience and outcomes analysis. Plast Reconstr Surg. 2011 Jan;127(1):173-180. doi: 10.1097/PRS.0b013e3181f95a36. PMID 21200211
- [Background] Bourke MJ, Hope RL, Chu G, Gillespie PE, Bull C, O'Rourke I, Williams SJ. Laser palliation of inoperable malignant dysphagia: initial and at death. Gastrointest Endosc. 1996 Jan;43(1):29-32. doi: 10.1016/s0016-5107(96)70256-0. PMID 8903814
- [Background] Briel JW, Tamhankar AP, Hagen JA, DeMeester SR, Johansson J, Choustoulakis E, Peters JH, Bremner CG, DeMeester TR. Prevalence and risk factors for ischemia, leak, and stricture of esophageal anastomosis: gastric pull-up versus colon interposition. J Am Coll Surg. 2004 Apr;198(4):536-41; discussion 541-2. doi: 10.1016/j.jamcollsurg.2003.11.026. PMID 15051003
- [Background] Buskens CJ, Hulscher JB, Fockens P, Obertop H, van Lanschot JJ. Benign tracheo-neo-esophageal fistulas after subtotal esophagectomy. Ann Thorac Surg. 2001 Jul;72(1):221-4. doi: 10.1016/s0003-4975(01)02701-1. PMID 11465183
- [Background] Collard JM, Tinton N, Malaise J, Romagnoli R, Otte JB, Kestens PJ. Esophageal replacement: gastric tube or whole stomach? Ann Thorac Surg. 1995 Aug;60(2):261-6; discussion 267. doi: 10.1016/0003-4975(95)00411-d. PMID 7646084
- [Background] D'Amico TA, Harpole DH Jr. Molecular biology of esophageal cancer. Chest Surg Clin N Am. 2000 Aug;10(3):451-69. PMID 10967750
- [Background] Domper Arnal MJ, Ferrandez Arenas A, Lanas Arbeloa A. Esophageal cancer: Risk factors, screening and endoscopic treatment in Western and Eastern countries. World J Gastroenterol. 2015 Jul 14;21(26):7933-43. doi: 10.3748/wjg.v21.i26.7933. PMID 26185366
- [Background] Edsander-Nord A, Jurell G, Wickman M. Donor-site morbidity after pedicled or free TRAM flap surgery: a prospective and objective study. Plast Reconstr Surg. 1998 Oct;102(5):1508-16. doi: 10.1097/00006534-199810000-00025. PMID 9774004
- [Background] El-Mrakby HH, Milner RH, McLean NR. Supercharged pedicled TRAM flap in breast reconstruction: is it a worthwhile procedure. Ann Plast Surg. 2002 Sep;49(3):252-7. doi: 10.1097/00000637-200209000-00003. PMID 12351972
- [Background] Ferguson A, Kingstone K. Coeliac disease and malignancies. Acta Paediatr Suppl. 1996 May;412:78-81. doi: 10.1111/j.1651-2227.1996.tb14259.x. PMID 8783767
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] Garcia-Vasquez C, Fernandez-Acenero MJ, Garcia Gomez-Heras S, Pastor C. Fibrin patch influences the expression of hypoxia-inducible factor-1alpha and nuclear factor-kappaBp65 factors on ischemic intestinal anastomosis. Exp Biol Med (Maywood). 2018 Jun;243(10):803-808. doi: 10.1177/1535370218777216. PMID 29932372
- [Background] GARLOCK JH. Resection of thoracic esophagus for carcinoma located above arch of aorta; cervical esophagogastrostomy. Surgery. 1948 Jul;24(1):1-8. No abstract available. PMID 18872828
- [Background] GARLOCK JH. Combined abdominothoracic approach for carcinoma of cardia and lower esophagus. Surg Gynecol Obstet. 1946 Dec;83(6):737-41. No abstract available. PMID 20275212
- [Background] Garvey PB, Buchel EW, Pockaj BA, Casey WJ 3rd, Gray RJ, Hernandez JL, Samson TD. DIEP and pedicled TRAM flaps: a comparison of outcomes. Plast Reconstr Surg. 2006 May;117(6):1711-9; discussion 1720-1. doi: 10.1097/01.prs.0000210679.77449.7d. PMID 16651940
- [Background] Goffi FS, Bevilacqua RG, Ferreira EA, Silva PA, Pinheiro Y, Lima EW, Bastos Eda S. [Surgery of cancer of he esophagus. Technic and results]. AMB Rev Assoc Med Bras. 1969 Jan;15(1):37-42. No abstract available. Portuguese. PMID 5306651
- [Background] Griffin SM, Lamb PJ, Dresner SM, Richardson DL, Hayes N. Diagnosis and management of a mediastinal leak following radical oesophagectomy. Br J Surg. 2001 Oct;88(10):1346-51. doi: 10.1046/j.0007-1323.2001.01918.x. PMID 11578290
- [Background] Grotting JC, Beckenstein MS, Arkoulakis NS. The art and science of autologous breast reconstruction. Breast J. 2003 Sep-Oct;9(5):350-60. doi: 10.1046/j.1524-4741.2003.09527.x. PMID 12968954
- [Background] Harashina T, Sone K, Inoue T, Fukuzumi S, Enomoto K. Augmentation of circulation of pedicled transverse rectus abdominis musculocutaneous flaps by microvascular surgery. Br J Plast Surg. 1987 Jul;40(4):367-70. doi: 10.1016/0007-1226(87)90039-7. PMID 2957016
- [Background] Scheflan M, Hartrampf CR, Black PW. Breast reconstruction with a transverse abdominal island flap. Plast Reconstr Surg. 1982 May;69(5):908-9. No abstract available. PMID 7071252
- [Background] Hermreck AS, Crawford DG. The esophageal anastomotic leak. Am J Surg. 1976 Dec;132(6):794-8. doi: 10.1016/0002-9610(76)90461-x. PMID 998871
- [Background] Holmstrom H. The free abdominoplasty flap and its use in breast reconstruction. An experimental study and clinical case report. Scand J Plast Reconstr Surg. 1979;13(3):423-27. doi: 10.3109/02844317909013092. PMID 396670
- [Background] Kassis ES, Kosinski AS, Ross P Jr, Koppes KE, Donahue JM, Daniel VC. Predictors of anastomotic leak after esophagectomy: an analysis of the society of thoracic surgeons general thoracic database. Ann Thorac Surg. 2013 Dec;96(6):1919-26. doi: 10.1016/j.athoracsur.2013.07.119. Epub 2013 Sep 24. PMID 24075499
- [Background] Kesler KA, Pillai ST, Birdas TJ, Rieger KM, Okereke IC, Ceppa D, Socas J, Starnes SL. "Supercharged" isoperistaltic colon interposition for long-segment esophageal reconstruction. Ann Thorac Surg. 2013 Apr;95(4):1162-8; discussion 1168-9. doi: 10.1016/j.athoracsur.2013.01.006. Epub 2013 Feb 21. PMID 23434255
- [Background] Kim EK, Lee TJ, Eom JS. Comparison of fat necrosis between zone II and zone III in pedicled transverse rectus abdominis musculocutaneous flaps: a prospective study of 400 consecutive cases. Ann Plast Surg. 2007 Sep;59(3):256-9. doi: 10.1097/01.sap.0000252770.15946.14. PMID 17721210
- [Background] Kim SH, Lee KS, Shim YM, Kim K, Yang PS, Kim TS. Esophageal resection: indications, techniques, and radiologic assessment. Radiographics. 2001 Sep-Oct;21(5):1119-37; discussion 1138-40. doi: 10.1148/radiographics.21.5.g01se031119. PMID 11553820
- [Background] Koop H. Gastroesophageal reflux disease and Barrett's esophagus. Endoscopy. 2004 Feb;36(2):103-9. doi: 10.1055/s-2004-814177. PMID 14765307
- [Background] Kroll SS. Bilateral breast reconstruction in very thin patients with extended free TRAM flaps. Br J Plast Surg. 1998 Oct;51(7):535-7. doi: 10.1054/bjps.1998.0014. PMID 9924407
- [Background] Lagergren J, Bergstrom R, Lindgren A, Nyren O. Symptomatic gastroesophageal reflux as a risk factor for esophageal adenocarcinoma. N Engl J Med. 1999 Mar 18;340(11):825-31. doi: 10.1056/NEJM199903183401101. PMID 10080844
- [Background] Lagergren J, Bergstrom R, Nyren O. Association between body mass and adenocarcinoma of the esophagus and gastric cardia. Ann Intern Med. 1999 Jun 1;130(11):883-90. doi: 10.7326/0003-4819-130-11-199906010-00003. PMID 10375336
- [Background] van Lanschot JJ, Hulscher JB, Buskens CJ, Tilanus HW, ten Kate FJ, Obertop H. Hospital volume and hospital mortality for esophagectomy. Cancer. 2001 Apr 15;91(8):1574-8. doi: 10.1002/1097-0142(20010415)91:83.0.co;2-2. PMID 11301408
- [Background] LONGMIRE WP Jr. A modification of the Roux technique for antethoracic esophageal reconstruction. Surgery. 1947 Jul;22(1):94-100. No abstract available. PMID 20249263
- [Background] Marck KW, van der Biezen JJ, Dol JA. Internal mammary artery and vein supercharge in TRAM flap breast reconstruction. Microsurgery. 1996;17(7):371-4. doi: 10.1002/(SICI)1098-2752(1996)17:73.0.CO;2-J. PMID 9379884
- [Background] Liebermann-Meffert DM, Meier R, Siewert JR. Vascular anatomy of the gastric tube used for esophageal reconstruction. Ann Thorac Surg. 1992 Dec;54(6):1110-5. doi: 10.1016/0003-4975(92)90077-h. PMID 1449294
- [Background] Morris SF, Taylor GI. Predicting the survival of experimental skin flaps with a knowledge of the vascular architecture. Plast Reconstr Surg. 1993 Dec;92(7):1352-61. PMID 8248411
- [Background] NAKAYAMA K. Statistical review of five-year survivals after surgery for carcinoma of the esophagus and cardiac portion of the stomach. Surgery. 1959 Jun;45(6):883-9. No abstract available. PMID 13659330
- [Background] Molina-Navarro C, Hosking SW, Hayward SJ, Flowerdew AD. Gastroaortic fistula as an early complication of esophagectomy. Ann Thorac Surg. 2001 Nov;72(5):1783-8. doi: 10.1016/s0003-4975(00)02569-8. PMID 11722100
- [Background] Pernia LR, Miller HL, Saltz R, Vasconez LO. "Supercharging" the rectus abdominis muscle to provide a single flap for cover of large mediastinal wound defects. Br J Plast Surg. 1991 May-Jun;44(4):243-6. doi: 10.1016/0007-1226(91)90064-q. PMID 2059779
- [Background] Rezai M, Darsow M, Kummel S, Kramer S. Autologous and alloplastic breast reconstruction--overview of techniques, indications and results. Gynakol Geburtshilfliche Rundsch. 2008;48(2):68-75. doi: 10.1159/000118934. Epub 2008 Apr 16. PMID 18431046
- [Background] Serletti JM. Breast reconstruction with the TRAM flap: pedicled and free. J Surg Oncol. 2006 Nov 1;94(6):532-7. doi: 10.1002/jso.20492. PMID 17061276
- [Background] Urschel JD. Ischemic conditioning of the stomach may reduce the incidence of esophagogastric anastomotic leaks complicating esophagectomy: a hypothesis. Dis Esophagus. 1997 Jul;10(3):217-9. doi: 10.1093/dote/10.3.217. PMID 9280083
- [Background] Valverde A, Hay JM, Fingerhut A, Elhadad A. Manual versus mechanical esophagogastric anastomosis after resection for carcinoma: a controlled trial. French Associations for Surgical Research. Surgery. 1996 Sep;120(3):476-83. doi: 10.1016/s0039-6060(96)80066-3. PMID 8784400
- [Background] Whooley BP, Law S, Murthy SC, Alexandrou A, Wong J. Analysis of reduced death and complication rates after esophageal resection. Ann Surg. 2001 Mar;233(3):338-44. doi: 10.1097/00000658-200103000-00006. PMID 11224620
- [Background] Yamamoto Y, Nohira K, Sugihara T, Shintomi Y, Ohura T. Superiority of the microvascularly augmented flap: analysis of 50 transverse rectus abdominis myocutaneous flaps for breast reconstruction. Plast Reconstr Surg. 1996 Jan;97(1):79-83; discussion 84-5. doi: 10.1097/00006534-199601000-00013. PMID 8532809